CLINICAL TRIAL: NCT06787339
Title: A Prospective, Single-arm,Clinical Trial Exploring the Efficacy and Safety of Chemotherapy De-escalation Using Capecitabine in Low-risk Early Triple-negative Breast Cancer
Brief Title: Capecitabine in Low Risk Triple Negative Breast Cancer
Acronym: Calorite
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N065
Record Dates: First submitted 2025-01-13; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy de-escalation; triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capecitabine (Experimental): capecitabine metronomic therapy for one year
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 650mg/m2, bid, p.o for 1 year

SUMMARY:
This study aims to evaluate the efficacy and safety of capecitabine as the only adjuvant chemotherapy drug in patients with low-risk early triple-negative breast cancer who have received adequate local treatment. Patients meeting the inclusion criteria will receive capecitabine metronomic therapy for one year.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of capecitabine as the only adjuvant chemotherapy drug in patients with low-risk T1N0M0 early triple-negative breast cancer who have received adequate local treatment. Patients meeting the inclusion criteria will receive capecitabine metronomic therapy for one year. The low-risk population defined in this study includes the IM subtype with abundant stromal tumor-infiltrating lymphocytes, or the LAR subtype with low ki-67 proliferation, or elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years;
2. Pathological confirmed of stage I breast cancer: histologically confirmed that the longest diameter of invasive cancer is no more than 2cm and the lymph node is negative (N0);
3. Histologically documented TNBC after early breast cancer surgery (absence of HER2, ER, and PR expression)
4. Patients who have undergone standard and adequate surgical treatment;
5. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN#and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula);
6. No evidence of metastasis in clinical or imaging examinations before surgery, that is, M0;
7. ECOG score of 0 or 1;
8. Meeting one of the low-risk criteria defined in this study: a) IM subtype, that is, the proportion of stromal tumor-infiltrating lymphocytes is high or CD8 is high; b) LAR subtype and ki-67 less than 20%; c) Age ≥ 70 years.

8)The patient voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy;
2. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ;
3. Has metastic (Stage 4) breast cancer;
4. Pregnant or breast feeding women, or people of childbearing age who cannot practice effective contraceptives;
5. Patients participating in other clinical trials at the same time;
6. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmHg, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension; Has severe or uncontrolled infection; 7) Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders; 8)The researchers considered patients to be unsuitable for the study. 9)Has bilateral breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
RFS | 3 years
  recurrence free survival

SECONDARY OUTCOMES:
iDFS | 3 years
  invasive disease-free survival
DRFS | 3 years
  distant relapse-free survival
DFS | 3 years
  disease-free survival
OS | 3 years
  overall survival
adverse events | 3 years
  adverse events according to CTCAE 5.0
PRO | 3 years
  patient reported outcome

CONTACTS AND LOCATIONS:
Locations (1):
- breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China